CLINICAL TRIAL: NCT05845905
Title: Effects of Remote Ischemic Conditioning on Blood Pressure in Older Patients With Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RICBP-HT
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Active Comparator): Patients are treated with remote ischemic conditioning (RIC).
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC group (Placebo Comparator): Patients are treated with sham remote ischemic conditioning (sham-RIC).
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by the inflation of an automated cuff to the pressure rising by 20 mmHg from baseline systolic pressure. RIC will be conducted twice daily for 7 days.
  Arms: RIC group
Procedure: Sham remote ischemic conditioning — Sham-RIC is performed in the same way as the treatment group except that the blood pressure cuff is inflated to 60 mmHg, which produces mild pressure sensations but has no blocking impact on blood flow.
  Arms: Sham RIC group

SUMMARY:
The purpose of this study is to learn about effects of remote ischemic conditioning on blood pressure in older patients with essential hypertension.

DETAILED DESCRIPTION:
Current studies have shown that remote ischemic conditioning can improve vascular endothelial function and inhibit sympathetic nervous system activity. Thus it may provide some organ protection as well as anti-hypertensive effects. The purpose of this study is to learn about effects of remote ischemic conditioning on blood pressure in older patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥65 years and ≤85 years, regardless of gender;
* 2) History of essential hypertension and clinical systolic blood pressure ≥ 140 mmHg, regardless of whether they are receiving antihypertensive medication;
* 3) Willing to participate and sign the informed consent.

Exclusion Criteria:

* 1) Secondary hypertension;
* 2) Clinical blood pressure ≥ 180/110 mmHg or 24-hour mean arterial pressure ≥ 170/100 mmHg;
* 3) Severe organ dysfunction or failure;
* 4) Severe hematologic disorders or significant coagulation abnormalities;
* 5) History of atrial fibrillation or myocardial infarction within 6 months;
* 6) Individuals who had contraindication of remote ischemic conditioning, such as severe soft tissue injury, fracture or vascular injury in the upper limb, acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
* 7) Individuals who will or have received anticoagulant therapy with drugs such as dabigatran, rivaroxaban, warfarin, etc;
* 8) Those who are participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to enrollment;
* 9) Other conditions that the researchers think are not suitable for the project.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean systolic blood pressure | 0-7 days
  Difference in mean value of systolic blood pressure during RIC/sham-RIC between two groups.

SECONDARY OUTCOMES:
Mean diastolic blood pressure | 0-7 days
  Difference in mean value of diastolic blood pressure during RIC/sham-RIC between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China